CLINICAL TRIAL: NCT04737811
Title: Validation and Reliability of the Turkish Translation of the Swallowing Disturbance Questionnaire in Parkinson's Disease Patients
Brief Title: Validation of the Turkish Swallowing Disturbance Questionnaire
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Sevgi Atar, Specialist, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 440
Record Dates: First submitted 2021-01-30; First posted 2021-02-04 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease; Dysphagia
Keywords: Parkinson's disease; dysphagia; questionnaire; swallowing; validation
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: The group consists of Parkinson's disease patients with dysphagia complaints. The participants will be given the Turkish version of the Swallow Disturbance Questionnaire (SDQ-T), which consisted of 15 questions and two scales evaluated with the fiberoptic endoscopic evaluation of swallowing. After two weeks, all participants will be given the SDQ-T for sampling.
  Interventions: Other: Turkish Version of Swallowing Disturbance Questionnaire

INTERVENTIONS:
Other: Turkish Version of Swallowing Disturbance Questionnaire — The Turkish Version of Swallowing Disturbance Questionnaire consists of 15 questions related with dysphagia.

SUMMARY:
Purpose of the study is the validity and reliability of the Turkish version of the Swallowing Disturbance Questionnaire (SDQ-T), so that it would be used as an assessment tool for Turkish Parkinson Disease's (PD) patients. Despite being translated and validated in many languages, there is no validated Turkish version of SDQ to measure the severity of dysphagia in PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) patients who suffered from dysphagia have reported significantly reduced quality of life. The swallow function is a multidirectional process that depends on complex neuro-muscular network. The function can be evaluated using instrumental, such as fibreoptic endoscopic evaluation of swallowing (FEES), videofluoroscopy, or well structured questionnaires. There are many questionnaire and scales for assessment of dysphagia in PD but very few have been validated. The study will assess the construct validity and reliability of the Turkish version of Swallowing Disturbance Questionnaire. The investigators developed the Turkish version of this questionnaire (SDQ-T), according to the cross-cultural adaptation guidelines. Two translators translated the SDQ into Turkish and a native English language speaker reverse-translated it into English. The back translation was sent to the original author for proofreading. The SDQ questionnaire consisted of 15 basic questions related with dysphagia symptoms in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease
* Able to speak, read, understand and write in Turkish
* Taking food orally
* Malignancy
* Having an active infection
* Advanced demans or

Exclusion Criteria:

* Diagnosed with other neurodegenerative disorders.
* Able not to speak, read, understand and write in Turkish
* Advanced demeans or other cognitive limitations
* Underwent any surgery last six months
* Pregnancy
* Underwent laryngectomy/neck dissection/tracheostomy/neck radiotherapy
* Out of age 18-80 years old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Turkish Version of Swallow Disturbance Questionnaire | Baseline
  Turkish version of the questionnaire consists of 15 questions about dysphagia and swallowing complaints. The minimum score is 0 and maximum score is 44,5. The lower scores mean a normal swallowing function, higher scores mean worst swallowing functions.
Turkish Version of Swallow Disturbance Questionnaire | 2 weeks
  Turkish version of the questionnaire consists of 15 questions about dysphagia and swallowing complaints. The minimum score is 0 and maximum score is 44,5. The lower scores mean a normal swallowing function, higher scores mean worst swallowing functions.
Penetration and aspiration scale | Baseline
  The scale consists of 8 levels for assessment of penetration and aspiration. The scores are from 0 to 8. Low score is better, higher score is worse.
Yale Pharyngeal Residue Severity Rating Scale | Baseline
  The scale consists of 5 assessment units and two localisations for pharyngeal residue. The scores are from 1 to 5 each localisation. Low score is better, higher score is worse.

SECONDARY OUTCOMES:
Subject demographics | Baseline
  The median values of age and ratio of gender in all groups

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Atar, Asso Prof,MD, Study Chair — University of Health Sciences, ENT Clinic, Prof Dr Cemil Tascioglu City Hospital; Sevgi Atar, Special.,MD, Study Director — University of Health Sciences, PMR Clinic, Prof Dr Cemil Tascioglu City Hospital; Onur Akan, Special.,MD, Principal Investigator — University of Health Sciences, Department of Neurology, Prof Dr Cemil Tascioglu City Hospital
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manor Y, Giladi N, Cohen A, Fliss DM, Cohen JT. Validation of a swallowing disturbance questionnaire for detecting dysphagia in patients with Parkinson's disease. Mov Disord. 2007 Oct 15;22(13):1917-21. doi: 10.1002/mds.21625. PMID 17588237
- [Background] Cohen JT, Manor Y. Swallowing disturbance questionnaire for detecting dysphagia. Laryngoscope. 2011 Jul;121(7):1383-7. doi: 10.1002/lary.21839. Epub 2011 Jun 10. PMID 21671239